CLINICAL TRIAL: NCT02673138
Title: Effect of Canagliflozin in T1DM After Interruption of Continuous Subcutaneous Insulin Infusion
Brief Title: Effect of Canagliflozin in T1DM (Type 1 Diabetes Melitus) After Interruption of Continuous Subcutaneous Insulin Infusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1508016333; 1K12DK094714-01 (NIH)
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2018-11-29 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-09

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Canagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Basal interruption (Active Comparator): Subjects will undergo basal interruption without canagliflozin during an overnight stay on the research unit
  Interventions: Other: basal interruption without canagliflozin
- Basal interruption with canagliflozin (Experimental): Subjects will undergo basal interruption with canagliflozin during an overnight stay on the research unit
  Interventions: Drug: canagliflozin

INTERVENTIONS:
Drug: canagliflozin — basal interruption with canagliflozin
  Other Names: Invokana
  Arms: Basal interruption with canagliflozin
Other: basal interruption without canagliflozin — basal interruption
  Arms: Basal interruption

SUMMARY:
This study will be an open-label, cross-over study as subjects will be studied under both study conditions - suspension of subcutaneous insulin infusion via pump during treatment with insulin alone (control) vs. suspension of subcutaneous insulin via pump during treatment with insulin and canagliflozin.

DETAILED DESCRIPTION:
The study will consist of 4 visits: an enrollment/screening visit, a control visit with pump suspension prior to treatment with canagliflozin, a visit with pump suspension while on canagliflozin and an end of study visit. Each of the pump suspension visits will be approximately 20-hour overnight admissions to the Hospital Research Unit (HRU).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 years
2. Clinical diagnosis of T1D (type 1 diabetes) (formal antibody and/or genetic testing will not be required)
3. Duration of T1D ≥ 1 year
4. HbA1c ≤ 9 %
5. Treated with continuous subcutaneous insulin infusion (with or without adjunctive treatment with a SGLT2 inhibitor) for at least 3 months
6. Body weight > 40 kg
7. Be in good general health without other acute or chronic illness that in the judgment of the investigator could interfere with the study or jeopardize subject safety
8. Normal hematocrit
9. Able to give consent
10. Female subjects of reproductive potential must be abstinent or consistently using appropriate family planning methods.

Exclusion Criteria:

1. Insulin resistant (defined as requiring > 1.5 units/kg/day at time of study enrollment)
2. Renal impairment, determined as eGFR < 60 ml/minute/1.73m2

   1. History of unstable or rapidly progressing renal disease
   2. Conditions of congenital renal glucosuria
   3. Renal allograft
   4. Recurrent UTI (urinary tract infection)
   5. History of Vesico-ureteral-reflux disease
3. Presence of any medical or psychiatric disorder that may interfere with subject safety or study conduct
4. Use of metformin, thiazolidinedione or GLP1 agonist within 1 month prior to screening visit. For those subjects on canagliflozin or other SGLT2 inhibitors, an alternate study procedure may be utilized as described above
5. Use of any medications (besides insulin or SGLT2 inhibitor) known to effect blood glucose levels, including oral or other systemic glucocorticoid therapy. Inhaled, intranasal, or rectal corticosteroid use is allowed as long as not given within 2 weeks of the closed loop admissions. Use of topical glucocorticoids is allowable as long as affected skin area does not overlap with study device sites
6. History of hypoglycemic seizure within last 3 months
7. History of diabetic ketoacidosis (DKA) requiring medical intervention (ie. emergency room visit and/or hospitalization) within 1 month prior to the screening visit
8. Allergies or contraindication to the contents of canagliflozin tablets or insulin
9. Volume depleted subjects. Subjects at risk for volume depletion due to co-existing conditions or concomitant medications, such as loop diuretics who cannot carefully monitor their volume status should be excluded from the study
10. Female subjects who are pregnant, lactating, or unwilling to be tested for pregnancy
11. Recurrent GU (genitourinary) infections
12. Uncircumcised males secondary to increased risk of development of GU infections
13. History of hypotension, defined as blood pressure (BP) <10th% for age and sex

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neha Patel, DO, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Basal Interruption With or Without Canagliflozin: Subjects will undergo basal interruption with or without canagliflozin during an overnight stay on the research unit
  canagliflozin: basal interruption with canagliflozin
Period: Overall Study
Arm/Group | Basal Interruption With or Without Canagliflozin
Started | 10
Started Day 1 | 10
Ended Day 1 | 10
Started Day 2 | 10
Ended Day 2 | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Basal Interruption With or Without Canagliflozin: Subjects will undergo basal interruption with canagliflozin during an overnight stay on the research unit
  canagliflozin: basal interruption with canagliflozin
Arm/Group | Basal Interruption With or Without Canagliflozin
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Differences in Plasma Glucose Levels Following the Interruption of Basal Subcutaneous Infusion of Insulin
Description: The primary outcome measure for this study will be differences in plasma glucose levels following the interruption of basal subcutaneous infusion of insulin under the two study conditions; i.e., control study during treatment with insulin alone vs. experimental study during treatment with insulin plus canagliflozin or other SGLT2 inhibitor.
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Basal Interruption | Basal Interruption With Canagliflozin
Number analyzed (Participants) | 10 | 10
mg/dL | 197 (24) | 99 (13)

2. Primary Outcome: Differences in BHB (Beta-hydroxybutyrate) Levels Following Interruption of Basal
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Basal Interruption | Basal Interruption With Canagliflozin
Number analyzed (Participants) | 10 | 10
mmol/L | 1.2 (0.2) | 1.5 (0.2)

3. Secondary Outcome: Differences in Free Fatty Acid Levels Following Interruption of Basal Subcutaneous Insulin Infusion
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: mmol/L
Arm/Group | Basal Interruption | Basal Interruption With Canagliflozin
Number analyzed (Participants) | 10 | 10
mmol/L | 0.8 (0.1) | 0.7 (0.1)

4. Secondary Outcome: Differences in Glucagon Levels Following the Interruption of the Basal Subcutaneous Insulin Infusion
Time Frame: 20 hours
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Basal Interruption | Basal Interruption With Canagliflozin
Number analyzed (Participants) | 10 | 10
pg/mL | 14 (5) | 36 (15)

ADVERSE EVENTS:
Arm/Group | Basal Interruption | Basal Interruption With Canagliflozin
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Basal Interruption (N=10) | Basal Interruption With Canagliflozin (N=10)
Vaginal Candidiasis (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes